CLINICAL TRIAL: NCT04749667
Title: Study of Mesenchymal Autologous Stem Cells as Regenerative Treatment for Multiple Sclerosis
Acronym: SMART-MS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other); University Hospital Ulm (Other); University Hospital, Akershus (Other); St. Olavs Hospital (Other); University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 159326
Record Dates: First submitted 2021-01-20; First posted 2021-02-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis; Progressive Multiple Sclerosis
Keywords: Mesenchymal stem cells; Multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, placebo-controlled, cross-over study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Crossover with MSCs at baseline and placebo at 6 months (Experimental): Receives mesenchymal stem cells at baseline and placebo at 6 months
  Interventions: Other: MSCs; Drug: Saline
- Arm B - Crossover with placebo at baseline and MSCs at 6 months (Experimental): Receives placebo at baseline and mesenchymal stem cells at 6 months
  Interventions: Other: MSCs; Drug: Saline

INTERVENTIONS:
Other: MSCs — Autologous bone-marrow derived mesenchymal stem cells
  Other Names: Mesenchymal stem cells
Drug: Saline — Isotonic saline

SUMMARY:
The primary objective of the study is to investigate neuroregenerative efficacy (proof of concept) of intrathecal treatment with autologous MSCs as measured by neurophysiological parameters in patients with progressive MS.

Secondary objectives are to assess neuroregenerative efficacy as measured by other neurophysiological parameters as well as clinical, opthalmological and MRI modalities, and to assess safety of the treatment procedure.

DETAILED DESCRIPTION:
Prospective, interventional, randomized, placebo-controlled, cross-over study. Patients are randomized to either treatment arm A or B.

Patients in both treatment arms receive intrathecal autologous MSCs, arm A at baseline and arm B at six months.

All patients undergo bone marrow (BM) aspiration prior to baseline. Patients in treatment arm A receive intrathecal autologous MSCs whereas patients in treatment arm B receive placebo. The treatment is blinded for the patients. The BM aspirate from patients in treatment arm B is processed, cryopreserved and stored in a biobank.

At six months, all patients undergo a second BM aspiration. Patients in treatment arm A now receive placebo. The BM aspirate from patients in treatment arm A is processed, cryopreserved and stored in a biobank. Patients in treatment arm B receive intrathecal autologous MSCs. The treatment is blinded for the patients.

Primary outcome is assessed at six months and secondary outcomes are assessed at six, twelve and eighteen months post baseline. Investigator assessing outcomes are blinded to patient treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 to ≤55, both genders
2. Diagnosis of secondary progressive or primary progressive MS using revised McDonald criteria of clinically definite MS
3. An EDSS score of 4 to 7
4. Disease duration 2 - 15 years
5. Signed, written informed consent

Exclusion Criteria:

1. Any illness or prior/ongoing treatment that in the opinion of the investigators would jeopardize the ability of the patient to tolerate autologous stem cell treatment
2. Any ongoing infection, including Tbc, CMV, EBV, HSV, VZV, hepatitis virus, toxoplasmosis, HIV or syphilis infections, as well as heaptitis B surface antigen positivity and/or hepatitis C PCR positivity
3. Current immunomodulatory/immunosuppressive treatment
4. Immunomodulatory/immunosuppressive treatment within 6 months prior to inclusion. This includes, but is not restricted to treatment with natalizumab, fingolimod, dimetylfumurat, glatiramer acetate, interferon beta medications, teriflunomide, and siponimod.
5. Treatment with kladribin, ocrelizumab, rituximab, and alemtuzumab within 12 months prior to inclusion
6. Treatment with hematopoietic stem cell therapy within 12 months prior to inclusion
7. Treatment with glucocorticoids or ACTH within three months prior to start of inclusion
8. Having experienced an MS relapse within 2 years prior to study inclusion
9. Current treatment with fampridin
10. History of malignancy other than basal cell carcinoma of the skin or carcinoma in situ that has been in remission for more than one year
11. Severely limited life expectancy by another co-morbid illness
12. History of previous diagnosis of myelodysplasia or previous hematologic disease (including lymphoproliferative disease, bone marrow insufficiency or previous lymphoid irradiation) or current clinically relevant abnormalities of white blood cell counts
13. Immunocompromised patients
14. Estimated glomerular filtration rate <60 ml/min/1.73 m2 or known renal failure
15. Bleeding or clotting diathesis or the use of antithrombotic or anticoagulative treatment
16. Platelet (thrombocyte) count <100 x 10*9/L
17. Participation in another experimental clinical study within the preceding 12 months
18. Contraindications to MRI
19. Prior or current major depression
20. Prior or current psychiatric illness, mental deficiency or cognitive dysfunction influencing the patient ability to make an informed consent or comply with the treatment and follow-up phases of this protocol.
21. Pregnancy or risk of pregnancy (this includes patients that are unwilling to practice active contraception during the duration of the study), breastfeeding or lactation
22. History of autologous/allogenic bone marrow transplantation or peripheral blood cell transplant
23. Known hypersensitivity against paracetamol, codein or xylocain
24. Diagnosis or strong suspicion of polyneuropathy
25. Prior or current alcohol or drug dependencies
26. Inability to give informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2024-10-04 (Estimated); Study Completion 2025-01-04 (Estimated)

PRIMARY OUTCOMES:
Neurophysiological parameters - Combined evoked potentials | 6 months
  Somatosensoric evoked potentials (SEP) + visual evoked potentials (VEP) + motor evoked potentials (MEP), latency (ms) and amplitude (mV)

SECONDARY OUTCOMES:
Neurophysiological parameters - Somatosensoric evoked potantials | 6 and 12 months
  SEP, latency (ms) and amplitude (mV)
Neurophysiological parameters - Motor evoked potentials | 6 and 12 months
  MEP, latency (ms) and amplitude (mV)
Neurophysiological parameters - Visual evoked potentials | 6 and 12 months
  VEP, latency (ms) and amplitude (mV)
MRI-Lesion volumes | 6 and 12 months
  T1- and T2-weighted hyperintense lesion volume
MR- Brain volumes | 6 and 12 months
  Brain volumes
Expanded disability status scale | 6, 12 and 18 months
  EDSS
Patient reported outcomes (PROs) | 6, 12 and 18 months
  Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS), European Quality of Life 5 dimensions (EQ-5D-5L), Multiple Sclerosis Impact Scale (MSIS) and Fatigue severity scale (FSS)
Nine-Hole-Peg Test (9-HPT) | 6, 12 and 18 months
  Nine-Hole-Peg Test (9-HPT)
Timed 25 Foot Walk (T25FW) | 6, 12 and 18 months
  Timed 25 Foot Walk (T25FW)
Visual function | 6, 12 and 18 months
  Visual acuity, visual field, color vision and contrast sensitivity
Optical coherence tomography (OCT) | 6, 12 and 18 months
  Retinal thickness
Rate and nature of adverse- and serious adverse events | 6, 12 and 18 months
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Elnan Kvistad, PhD, Principal Investigator — Haukeland University Hospital; Lars Bø, Prof, Study Chair — Haukeland University Hospital
Locations (4):
- Norway (4):
  - Akershus university hospital, Lørenskog, Akershus
  - University hospital of North Norway, Tromsø, Troms Og Finnmark
  - St.Olav university hospital, Trondheim, Trøndelag
  - Haukeland University Hospital, Bergen, Vestland